CLINICAL TRIAL: NCT06427005
Title: Fruquintinib Combined with S-1 and Raltitrexed for Patients with Metastatic Colorectal Cancer Refractory to Standard Therapies: a Phase II Study
Brief Title: Fruquintinib Plus S-1 and Raltitrexed (RSF) for MCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Meng Qiu (Other)
Collaborators: Beijing Xisike Clinical Oncology Research Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Meng Qiu, Principal Investigator, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-71
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-05

CONDITIONS: Fruquintinib; S-1; Raltitrexed
Keywords: S-1; Fruquintinib; raltitrexed
MeSH Terms: interventions — HMPL-013; S 1 (combination); Tegafur; gimeracil; potassium oxonate; raltitrexed

STUDY DESIGN:
Intervention Model Description: Participants received Fruquintinib (5 mg daily for 14 days followed by a 7-day break), oral S-1 (80-120 mg daily for 14 days, followed by a 7-day break), and raltitrexed (3 mg/m² on day 1, with a maximum dose of 5 mg) every 3 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RSF treatment arm (Experimental): Participants received Fruquintinib (5 mg daily for 14 days followed by a 7-day break), oral S-1 (80-120 mg daily for 14 days, followed by a 7-day break), and raltitrexed (3 mg/m² on day 1, with a maximum dose of 5 mg) every 3 weeks.
  Interventions: Drug: Fruquintinib; Drug: S-1; Drug: raltitrexed

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib 5 mg daily for 14 days followed by a 7-day break
  Other Names: Elunate
Drug: S-1 — S-1 80-120 mg daily for 14 days, followed by a 7-day break
  Other Names: Tegafur,Gimeracil and Oteracil Potassium Capsules
Drug: raltitrexed — raltitrexed 3 mg/m² on day 1, with a maximum dose of 5 mg
  Other Names: thymidylate synthase inhibitor

SUMMARY:
Based on the FRECO-2 study, Fruquintinib has become one of the standard third-line treatments for advanced colorectal cancer; however, its objective response rate (ORR) remains low. Our previous studies have shown that the combination of raltitrexed and S-1 -/+ bevacizumab is effective and provides a significant survival benefit in patients with metastatic colorectal cancer (mCRC) who are refractory to standard treatments. This study aims to evaluate the efficacy and safety of combining Fruquintinib with S-1 and raltitrexed in these patients.

DETAILED DESCRIPTION:
Conducted at West China Hospital in China, this investigator-initiated, open-label, single-arm, phase II trial included patients with mCRC that had progressed following treatment with fluoropyrimidine, irinotecan, and oxaliplatin, and had at least one measurable lesion. Patients could have previously received anti-EGFR (for tumors with wild-type RAS) and anti-VEGF therapy in the first or second line, including those who had been treated with bevacizumab in two consecutive chemotherapy regimens. Participants received Fruquintinib (5 mg daily for 14 days followed by a 7-day break), oral S-1 (80-120 mg daily for 14 days, followed by a 7-day break), and raltitrexed (3 mg/m² on day 1, with a maximum dose of 5 mg) every 3 weeks. The primary endpoint was the ORR, while secondary endpoints included progression-free survival (PFS), overall survival (OS), and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, any gender.
2. Patients with metastatic colorectal adenocarcinoma confirmed by pathological histology or cytology.
3. Expected survival time ≥ 12 weeks.
4. ECOG score of 0-2.
5. Previously treated for metastatic colorectal cancer with fluoropyrimidine (allowing intravenous and/or oral fluoropyrimidine formulations, excluding DPD enzyme inhibitors), irinotecan, and oxaliplatin chemotherapy, which failed (treatment failure defined as intolerable adverse reactions, disease progression during treatment, or disease progression within 6 months after completing adjuvant chemotherapy); regardless of prior use of targeted drugs such as cetuximab or bevacizumab.
6. Patients must have an interval of at least 2 weeks since the last chemotherapy (at least 1 week for oral chemotherapy drugs) or more than 4 weeks since the end of radiotherapy, with the study's observable lesions located outside the radiotherapy target area.
7. According to RECIST 1.1 criteria, at least one measurable tumor lesion with a maximum diameter ≥ 1 cm as determined by spiral CT scan.
8. Laboratory test results within 1 week before enrollment must meet the following criteria:

   1. Hemoglobin ≥ 90 g/L; Platelets (PLT) ≥ 75 × 10^9/L;
   2. White blood cells (WBC) ≥ 3.0 × 10^9/L; Neutrophils (ANC) ≥ 1.5 × 10^9/L;
   3. Serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN);
   4. Total bilirubin (TBI) ≤ 1.5 × ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN if there is liver metastasis).
9. No prior use of raltitrexed or S-1 (or DPD enzyme inhibitors) in the treatment of colorectal cancer.
10. Signed informed consent.

Exclusion Criteria:

1. Patients unable to take oral medications.
2. Patients who have previously been treated with small molecule TKI drugs.
3. Patients with severe hepatic or renal insufficiency, or a recent history of myocardial infarction (within 3 months).
4. Patients with a history of other malignancies within the past five years, except for cured cervical carcinoma in situ and basal cell carcinoma of the skin.
5. Patients with a history of inflammatory bowel disease or extensive colonic resection, ≥50% or extensive small bowel resection with chronic diarrhea, or intestinal obstruction.
6. Patients with severe uncontrolled internal medical conditions or acute infections (fever > 38°C due to infection).
7. Patients with symptomatic brain or leptomeningeal metastases (unless the patient has been treated for brain or leptomeningeal metastases > 6 months, with negative imaging results within 4 weeks before study entry, and has stable clinical symptoms related to brain or leptomeningeal metastases at study entry).
8. Patients with clinically significant, uncontrolled pleural effusion or ascites despite clinical intervention.
9. Pregnant or breastfeeding women, or patients of reproductive potential (males or females not in menopause for less than 1 year) unwilling to use contraception.
10. Patients known to be allergic to raltitrexed, S-1, and Fruquintinib or any of their components.
11. Patients deemed unsuitable for participation in this clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
ORR | about a year
  Objective Response Rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version. 1.1

SECONDARY OUTCOMES:
DCR | about a year
  Disease Control Rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version. 1.1
OS | about a year
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up
Safety and tolerability | about a year
  Version 5.0 and AEs leading to dose interruption or discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Qiu, MD., Study Director — Sichuan University
Locations (2):
- China (2):
  - Sichuan University West China Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leng W, Wen Z, Wang H, Cao P, Liu J, Luo D, Qiu M. Raltitrexed, S-1 and fruquintinib (RSF) in the treatment of refractory metastatic colorectal cancer: study protocol for a multicenter, prospective, single-arm, phase II trial. BMC Cancer. 2025 Feb 28;25(1):376. doi: 10.1186/s12885-025-13654-7. PMID 40022044